CLINICAL TRIAL: NCT03033745
Title: An Open-label Multicenter Study to Evaluate the Safety and Tolerability of Higher Infusion Parameters of Immune Globulin Subcutaneous (Human), 20% Liquid (Hizentra®) in Subjects With Primary Immunodeficiency
Brief Title: Safety and Tolerability of Higher Infusion Parameters of IgPro20 (Hizentra) in Subjects With Primary Immunodeficiency (PID)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IgPro20_4004; 2016-003799-33 (EudraCT Number)
Record Dates: First submitted 2017-01-23; First posted 2017-01-27 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IgPro20 (Pump-Assisted Volume Cohort) (Experimental): Weekly volumes per injection site of 25 mL up to 50 mL administered subcutaneously.
  Interventions: Drug: IgPro20
- IgPro20 (Pump Assisted Flow Rate Cohort) (Experimental): Weekly flow rates per injection site of 25 mL/hour up to 100 mL/hour administered subcutaneously.
  Interventions: Drug: IgPro20
- IgPro20 (Manual Push Flow Rate Cohort) (Experimental): Frequent (ie, 2 to 7 times per week) flow rates per injection site of 25 to 30 mL/hour up to 120 mL/hour (equivalent of approximately 0.5 mL/minute up to 2 mL/minute) administered subcutaneously.
  Interventions: Drug: IgPro20

INTERVENTIONS:
Drug: IgPro20 — A liquid formulation of normal human IgG at a concentration of 20% administered as a subcutaneous infusion at a dose prescribed by subject's physician prior to study entry.
  Other Names: Hizentra

SUMMARY:
This multicenter, open-label, parallel-arm, non-randomized study is designed to evaluate safety and tolerability of higher infusion parameters of IgPro20 in subjects with primary immunodeficiency (PID). A total of 45 subjects (including at least 14 [30%] pediatric subjects ≤ 17 years of age and at least 9 [20%] obese subjects with body mass index [BMI] of ≥30 kg/m2) with confirmed PID will be evaluated in the study. The study will include three cohorts of 15 subjects each as follows: i) Pump-Assisted Volume Cohort (weekly infusions), volume per injection site of 25 mL up to 50 mL, ii) Pump Assisted Flow Rate Cohort (weekly infusions), flow rate per injection site of 25 mL/hour up to 100 mL/hour, iii) Manual Push Flow Rate Cohort (2 to 7 infusions per week), flow rate per injection site of 25 to 30 mL/hour up to 120 mL/hour (equivalent of approximately 0.5 mL/minute up to 2 mL/minute). Each cohort will test 3 infusion parameter levels (4 for the pump-assisted flow rate cohort), repeated at least 4 times over a duration of 12 weeks (16 weeks for the flow rate cohort). After 4 infusion weeks at each level, qualifying subjects (responders) will switch to the next infusion parameter level (eg, from 25 to 50 mL/h). During the study, the weekly dose will remain unchanged (as prescribed by treating physician, usually within 100-200 mg/kg per week range); only the respective infusion parameter under evaluation will change.

ELIGIBILITY:
Inclusion Criteria:

* Male or female on stable dose of IgPro20 (Hizentra) therapy.
* Women of childbearing potential must be using and agree to continue using medically approved contraception (which must be discussed with the study doctor) and must have a negative pregnancy test at screening.
* Subjects with PID, eg, with a diagnosis of common variable immunodeficiency or X-linked agammaglobulinemia, as defined by the Pan American Group for Immune Deficiency and the European Society of Immune Deficiencies.
* With infusion parameters as specified below:

Pump-Assisted Flow Rate Cohort subjects only

* Experience with pump-assisted infusions of IgPro20 at the tolerated flow rate of 25 mL/h per injection site for at least 1 month prior to Day 1.

Pump-Assisted Volume Cohort subjects only

* Total weekly IgPro20 dose of ≥ 50 mL (≥ 10 g).
* Experience with pump-assisted infusions of IgPro20 at tolerated volumes of 25 mL/injection site for at least 1 month prior to Day 1.

Manual Push Flow Rate Cohort subjects only

* Experience with frequent (2-7 times per week) infusions of IgPro20 at the tolerated flow rate of approximately 0.5 mL/min (equivalent of 25-30 mL/h) per injection site for at least 1 month prior to Day 1. The dose (volume) per injection site should not exceed 25 mL.

Exclusion Criteria:

* Ongoing serious bacterial infections at the time of screening.
* Other significant medical conditions that could increase the risk to the subject.
* Females who are pregnant, breast feeding, or planning a pregnancy during the course study.
* Participation in a study with an Investigational Medicinal Product (IMP) other than IgPro20 within three months prior to enrollment.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — CSL Behring
Locations (12):
- United States (10):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - University of Southern Florida, St. Petersburg, Florida
  - Georgia Pollens Clinical Research Centers, Albany, Georgia
  - Long Island Jewish Medical Center, Great Neck, New York
  - Icahn Medical Institute, New York, New York
  - Center for Clinical Research Rochester General Hospital, Rochester, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson JT, Bonagura VR, Cowan J, Hsu C, Mustafa SS, Patel NC, Routes JM, Sriaroon P, Vinh DC, Hofmann JH, Praus M, Rojavin MA. Safety and Tolerability of Subcutaneous IgPro20 at High Infusion Parameters in Patients with Primary Immunodeficiency: Findings from the Pump-Assisted Administration Cohorts of the HILO Study. J Clin Immunol. 2021 Feb;41(2):458-469. doi: 10.1007/s10875-020-00912-5. Epub 2021 Jan 6. PMID 33409867
- [Derived] Cowan J, Bonagura VR, Lugar PL, Maglione PJ, Patel NC, Vinh DC, Hofmann JH, Praus M, Rojavin MA. Safety and Tolerability of Manual Push Administration of Subcutaneous IgPro20 at High Infusion Rates in Patients with Primary Immunodeficiency: Findings from the Manual Push Administration Cohort of the HILO Study. J Clin Immunol. 2021 Jan;41(1):66-75. doi: 10.1007/s10875-020-00876-6. Epub 2020 Oct 6. PMID 33025378

RESULTS

PARTICIPANT FLOW:
Groups:
- IgPro20 (Pump-Assisted Volume Cohort): Volumes per injection site of 25 mL up to 50 mL administered subcutaneously.
  IgPro20: A liquid formulation of normal human IgG at a concentration of 20% administered as a weekly subcutaneous infusion at a dose prescribed by subject's physician prior to study entry.
- IgPro20 (Pump Assisted Flow Rate Cohort): Flow rates per injection site of 25 mL/hour up to 100 mL/hour administered subcutaneously.
  IgPro20: A liquid formulation of normal human IgG at a concentration of 20% administered as a weekly subcutaneous infusion at a dose prescribed by subject's physician prior to study entry.
- IgPro20 (Manual Push Flow Rate Cohort): Frequent infusions per week (2 to 7 times) with flow rates per injection site of approximately 25 to 30 mL/hour up to approximately 120 mL/hour (equivalent of approximately 0.5 mL/minute up to 2 mL/minute) administered subcutaneously.
  IgPro20: A liquid formulation of normal human IgG at a concentration of 20% administered as a subcutaneous infusion at a dose prescribed by subject's physician prior to study entry.
Period: Overall Study
Arm/Group | IgPro20 (Pump-Assisted Volume Cohort) | IgPro20 (Pump Assisted Flow Rate Cohort) | IgPro20 (Manual Push Flow Rate Cohort)
Started | 15 | 18 | 16
Completed | 14 | 17 | 14
Not Completed | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IgPro20 (Pump-Assisted Volume Cohort) | IgPro20 (Pump Assisted Flow Rate Cohort) | IgPro20 (Manual Push Flow Rate Cohort) | Total
Number analyzed (Participants) | 15 | 18 | 16 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 11 | 1 | 12
  Between 18 and 65 years | 14 | 5 | 14 | 33
  >=65 years | 1 | 2 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (14.18) | 26.7 (24.52) | 47.9 (13.28) | 40.5 (20.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 10 | 29
  Male | 6 | 8 | 6 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 14 | 16 | 12 | 42
  More than one race | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 0 | 6 | 9
  United States | 12 | 18 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders
Description: A responder is a subject within the Pump-Assisted Cohorts that performs at least 3 out of 4 valid infusions at a certain infusion parameter level (weekly volumes per injection site of 25-50 mL; weekly flow rates per injection site of 25-100 mL/hour). Determination of a responder in the Manual Push Cohort is more complex due to the expected variable frequency of infusions per week (ie, 5-17) for different subjects. A responder within the Manual Push Cohort is a subject that performs a minimum number of valid infusions during 4 weeks corresponding to a certain flow rate level ([ie, 2-7 times per week], flow rates per injection site of 30-120 mL/hour). Valid infusions do not need to be consecutive, but each subject needs to adhere to the same schedule (number of infusions per week) throughout the study. An infusion parameter will be considered successful if at least one third (≥ 33%) of the subjects in the corresponding cohort are responders at that infusion parameter level.
Time Frame: At the end of 4 weeks for each planned infusion parameter
Population: The Safety Analysis Set (SAS) comprised all subjects in the Full Analysis Set who received ≥ 1 dose or a partial dose of IgPro20 in the study.
Measure: Number; unit: percentage of responders
Arm/Group | IgPro20 (Pump-Assisted Volume Cohort) | IgPro20 (Pump Assisted Flow Rate Cohort) | IgPro20 (Manual Push Flow Rate Cohort)
Number analyzed (Participants) | 15 | 18 | 16
percentage of responders
  25 ml: number analyzed (Participants) | 15 | 0 | 0
  25 ml | 86.7 |  |
  40 ml: number analyzed (Participants) | 15 | 0 | 0
  40 ml | 73.3 |  |
  50 ml: number analyzed (Participants) | 15 | 0 | 0
  50 ml | 73.3 |  |
  25 ml/h: number analyzed (Participants) | 0 | 18 | 0
  25 ml/h |  | 77.8 |
  50 ml/h: number analyzed (Participants) | 0 | 18 | 0
  50 ml/h |  | 77.8 |
  75 ml/h: number analyzed (Participants) | 0 | 18 | 0
  75 ml/h |  | 66.7 |
  100 ml/h: number analyzed (Participants) | 0 | 18 | 0
  100 ml/h |  | 61.1 |
  30 ml/h: number analyzed (Participants) | 0 | 0 | 16
  30 ml/h |  |  | 100.0
  60 ml/h: number analyzed (Participants) | 0 | 0 | 16
  60 ml/h |  |  | 100.0
  120 ml/h: number analyzed (Participants) | 0 | 0 | 16
  120 ml/h |  |  | 87.5

2. Secondary Outcome: Rate of Treatment-emergent Adverse Events (TEAEs) Per Infusion
Description: Adverse event rate per infusion = number of adverse events/total number of infusions prior to subject's start date of non-response. Only events are included which start prior to subject's start date of non-response.
Time Frame: At the end of 4 weeks for each planned infusion parameter
Population: SAS
Measure: Number; unit: Number of TEAEs/infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro20 (Pump-Assisted Volume Cohort) | IgPro20 (Pump Assisted Flow Rate Cohort) | IgPro20 (Manual Push Flow Rate Cohort)
Number analyzed (Participants) | 15 | 18 | 16
Number analyzed (Infusions) | 152 | 222 | 626
Number of TEAEs/infusion
  25 ml: number analyzed (Participants) | 15 | 0 | 0
  25 ml: number analyzed (Infusions) | 60 | 0 | 0
  25 ml | 0.183 |  |
  40 ml: number analyzed (Participants) | 12 | 0 | 0
  40 ml: number analyzed (Infusions) | 48 | 0 | 0
  40 ml | 0.188 |  |
  50 ml: number analyzed (Participants) | 11 | 0 | 0
  50 ml: number analyzed (Infusions) | 44 | 0 | 0
  50 ml | 0.023 |  |
  25 ml/h: number analyzed (Participants) | 0 | 18 | 0
  25 ml/h: number analyzed (Infusions) | 0 | 70 | 0
  25 ml/h |  | 0.329 |
  50 ml/h: number analyzed (Participants) | 0 | 14 | 0
  50 ml/h: number analyzed (Infusions) | 0 | 55 | 0
  50 ml/h |  | 0.255 |
  75 ml/h: number analyzed (Participants) | 0 | 13 | 0
  75 ml/h: number analyzed (Infusions) | 0 | 50 | 0
  75 ml/h |  | 0.140 |
  100 ml/h: number analyzed (Participants) | 0 | 12 | 0
  100 ml/h: number analyzed (Infusions) | 0 | 47 | 0
  100 ml/h |  | 0.085 |
  30 ml/h: number analyzed (Participants) | 0 | 0 | 16
  30 ml/h: number analyzed (Infusions) | 0 | 0 | 220
  30 ml/h |  |  | 0.064
  60 ml/h: number analyzed (Participants) | 0 | 0 | 16
  60 ml/h: number analyzed (Infusions) | 0 | 0 | 208
  60 ml/h |  |  | 0.111
  120 ml/h: number analyzed (Participants) | 0 | 0 | 14
  120 ml/h: number analyzed (Infusions) | 0 | 0 | 198
  120 ml/h |  |  | 0.081

3. Secondary Outcome: Rate of Local TEAEs Per Infusion
Description: Local adverse event rate per infusion = number of local adverse events/total number of infusions prior to subject's start date of non-response. Local Adverse Events: comprises all events reported within the MedDRA high level terms "administration site reactions NEC (Not Elsewhere Classified)", "infusion site reactions", and "injection site reactions". Only events are included which start prior to subject's start date of non-response.
Time Frame: At the end of 4 weeks for each planned infusion parameter
Population: SAS
Measure: Number; unit: Number of local TEAEs/infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro20 (Pump-Assisted Volume Cohort) | IgPro20 (Pump Assisted Flow Rate Cohort) | IgPro20 (Manual Push Flow Rate Cohort)
Number analyzed (Participants) | 15 | 18 | 16
Number analyzed (Infusions) | 152 | 222 | 626
Number of local TEAEs/infusion
  25 ml: number analyzed (Participants) | 15 | 0 | 0
  25 ml: number analyzed (Infusions) | 60 | 0 | 0
  25 ml | 0.150 |  |
  40 ml: number analyzed (Participants) | 12 | 0 | 0
  40 ml: number analyzed (Infusions) | 48 | 0 | 0
  40 ml | 0.063 |  |
  50 ml: number analyzed (Participants) | 11 | 0 | 0
  50 ml: number analyzed (Infusions) | 44 | 0 | 0
  50 ml | 0.0 |  |
  25 ml/h: number analyzed (Participants) | 0 | 18 | 0
  25 ml/h: number analyzed (Infusions) | 0 | 70 | 0
  25 ml/h |  | 0.286 |
  50 ml/h: number analyzed (Participants) | 0 | 14 | 0
  50 ml/h: number analyzed (Infusions) | 0 | 55 | 0
  50 ml/h |  | 0.145 |
  75 ml/h: number analyzed (Participants) | 0 | 13 | 0
  75 ml/h: number analyzed (Infusions) | 0 | 50 | 0
  75 ml/h |  | 0.040 |
  100 ml/h: number analyzed (Participants) | 0 | 12 | 0
  100 ml/h: number analyzed (Infusions) | 0 | 47 | 0
  100 ml/h |  | 0.021 |
  30 ml/h: number analyzed (Participants) | 0 | 0 | 16
  30 ml/h: number analyzed (Infusions) | 0 | 0 | 220
  30 ml/h |  |  | 0.027
  60 ml/h: number analyzed (Participants) | 0 | 0 | 16
  60 ml/h: number analyzed (Infusions) | 0 | 0 | 208
  60 ml/h |  |  | 0.082
  120 ml/h: number analyzed (Participants) | 0 | 0 | 14
  120 ml/h: number analyzed (Infusions) | 0 | 0 | 198
  120 ml/h |  |  | 0.025

4. Secondary Outcome: Time to Onset of Local TEAEs
Description: Local Adverse Events: comprises all events reported within the MedDRA high level terms "administration site reactions NEC", "infusion site reactions", and "injection site reactions". Only events are included which start prior to subject's start date of non-response.
Time Frame: At the end of 4 weeks for each planned infusion parameter
Population: SAS
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Local TEAEs
Arm/Group | IgPro20 (Pump-Assisted Volume Cohort) | IgPro20 (Pump Assisted Flow Rate Cohort) | IgPro20 (Manual Push Flow Rate Cohort)
Number analyzed (Participants) | 15 | 18 | 16
Number analyzed (Local TEAEs) | 12 | 31 | 28
Days
  25 ml: number analyzed (Participants) | 15 | 0 | 0
  25 ml: number analyzed (Local TEAEs) | 9 | 0 | 0
  25 ml | 1.3 (2.45) |  |
  40 ml: number analyzed (Participants) | 12 | 0 | 0
  40 ml: number analyzed (Local TEAEs) | 3 | 0 | 0
  40 ml | 0 (0.0) |  |
  50 ml: number analyzed (Participants) | 11 | 0 | 0
  50 ml: number analyzed (Local TEAEs) | 0 | 0 | 0
  25 ml/h: number analyzed (Participants) | 0 | 18 | 0
  25 ml/h: number analyzed (Local TEAEs) | 0 | 20 | 0
  25 ml/h |  | 1.7 (2.94) |
  50 ml/h: number analyzed (Participants) | 0 | 14 | 0
  50 ml/h: number analyzed (Local TEAEs) | 0 | 8 | 0
  50 ml/h |  | 0.0 (0.04) |
  75 ml/h: number analyzed (Participants) | 0 | 13 | 0
  75 ml/h: number analyzed (Local TEAEs) | 0 | 2 | 0
  75 ml/h |  | 0 (0.0) |
  100 ml/h: number analyzed (Participants) | 0 | 12 | 0
  100 ml/h: number analyzed (Local TEAEs) | 0 | 1 | 0
  100 ml/h |  | 0 (NA) — Not estimable because events = 1 |
  30 ml/h: number analyzed (Participants) | 0 | 0 | 16
  30 ml/h: number analyzed (Local TEAEs) | 0 | 0 | 6
  30 ml/h |  |  | 0.2 (0.41)
  60 ml/h: number analyzed (Participants) | 0 | 0 | 16
  60 ml/h: number analyzed (Local TEAEs) | 0 | 0 | 17
  60 ml/h |  |  | 0.3 (0.59)
  120 ml/h: number analyzed (Participants) | 0 | 0 | 14
  120 ml/h: number analyzed (Local TEAEs) | 0 | 0 | 5
  120 ml/h |  |  | 0.2 (0.45)

5. Secondary Outcome: Intensity of Local TEAEs
Description: Mild = A type of AE that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. Moderate = A type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the subject. Severe = A type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Only events are included which start prior to subject's start date of non-response.
Time Frame: At the end of 4 weeks for each planned infusion parameter
Population: SAS
Measure: Count of Participants; unit: Participants
Arm/Group | IgPro20 (Pump-Assisted Volume Cohort) | IgPro20 (Pump Assisted Flow Rate Cohort) | IgPro20 (Manual Push Flow Rate Cohort)
Number analyzed (Participants) | 15 | 18 | 16
Participants
  25 ml (mild): number analyzed (Participants) | 15 | 0 | 0
  25 ml (mild) | 3 |  |
  25 ml (moderate): number analyzed (Participants) | 15 | 0 | 0
  25 ml (moderate) | 0 |  |
  25 ml (severe): number analyzed (Participants) | 15 | 0 | 0
  25 ml (severe) | 0 |  |
  40 ml (mild): number analyzed (Participants) | 12 | 0 | 0
  40 ml (mild) | 1 |  |
  40 ml (moderate): number analyzed (Participants) | 12 | 0 | 0
  40 ml (moderate) | 0 |  |
  40 ml (severe): number analyzed (Participants) | 12 | 0 | 0
  40 ml (severe) | 0 |  |
  50 ml (mild): number analyzed (Participants) | 11 | 0 | 0
  50 ml (mild) | 0 |  |
  50 ml (moderate): number analyzed (Participants) | 11 | 0 | 0
  50 ml (moderate) | 0 |  |
  50 ml (severe): number analyzed (Participants) | 11 | 0 | 0
  50 ml (severe) | 0 |  |
  25 ml/h (mild): number analyzed (Participants) | 0 | 18 | 0
  25 ml/h (mild) |  | 4 |
  25 ml/h (moderate): number analyzed (Participants) | 0 | 18 | 0
  25 ml/h (moderate) |  | 2 |
  25 ml/h (severe): number analyzed (Participants) | 0 | 18 | 0
  25 ml/h (severe) |  | 0 |
  50 ml/h (mild): number analyzed (Participants) | 0 | 14 | 0
  50 ml/h (mild) |  | 3 |
  50 ml/h (moderate): number analyzed (Participants) | 0 | 14 | 0
  50 ml/h (moderate) |  | 0 |
  50 ml/h (severe): number analyzed (Participants) | 0 | 14 | 0
  50 ml/h (severe) |  | 0 |
  75 ml/h (mild): number analyzed (Participants) | 0 | 13 | 0
  75 ml/h (mild) |  | 1 |
  75 ml/h (moderate): number analyzed (Participants) | 0 | 13 | 0
  75 ml/h (moderate) |  | 0 |
  75 ml/h (severe): number analyzed (Participants) | 0 | 13 | 0
  75 ml/h (severe) |  | 0 |
  100 ml/h (mild): number analyzed (Participants) | 0 | 12 | 0
  100 ml/h (mild) |  | 0 |
  100 ml/h (moderate): number analyzed (Participants) | 0 | 12 | 0
  100 ml/h (moderate) |  | 0 |
  100 ml/h (severe): number analyzed (Participants) | 0 | 12 | 0
  100 ml/h (severe) |  | 1 |
  30 ml/h (mild): number analyzed (Participants) | 0 | 0 | 16
  30 ml/h (mild) |  |  | 3
  30 ml/h (moderate): number analyzed (Participants) | 0 | 0 | 16
  30 ml/h (moderate) |  |  | 0
  30 ml/h (severe): number analyzed (Participants) | 0 | 0 | 16
  30 ml/h (severe) |  |  | 0
  60 ml/h (mild): number analyzed (Participants) | 0 | 0 | 16
  60 ml/h (mild) |  |  | 4
  60 ml/h (moderate): number analyzed (Participants) | 0 | 0 | 16
  60 ml/h (moderate) |  |  | 0
  60 ml/h (severe): number analyzed (Participants) | 0 | 0 | 16
  60 ml/h (severe) |  |  | 0
  120 ml/h (mild): number analyzed (Participants) | 0 | 0 | 14
  120 ml/h (mild) |  |  | 2
  120 ml/h (moderate): number analyzed (Participants) | 0 | 0 | 14
  120 ml/h (moderate) |  |  | 0
  120 ml/h (severe): number analyzed (Participants) | 0 | 0 | 14
  120 ml/h (severe) |  |  | 0

6. Secondary Outcome: Duration of Local TEAEs
Description: Local Adverse Events: comprises all events reported within the MedDRA high level terms "administration site reactions NEC", "infusion site reactions", and "injection site reactions".
Time Frame: At the end of 4 weeks for each planned infusion parameter
Population: SAS
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Local TEAEs
Arm/Group | IgPro20 (Pump-Assisted Volume Cohort) | IgPro20 (Pump Assisted Flow Rate Cohort) | IgPro20 (Manual Push Flow Rate Cohort)
Number analyzed (Participants) | 15 | 18 | 16
Number analyzed (Local TEAEs) | 12 | 31 | 28
Days
  25 ml: number analyzed (Participants) | 15 | 0 | 0
  25 ml: number analyzed (Local TEAEs) | 9 | 0 | 0
  25 ml | 2.2 (1.30) |  |
  40 ml: number analyzed (Participants) | 12 | 0 | 0
  40 ml: number analyzed (Local TEAEs) | 3 | 0 | 0
  40 ml | 2.7 (2.08) |  |
  50 ml: number analyzed (Participants) | 11 | 0 | 0
  50 ml: number analyzed (Local TEAEs) | 0 | 0 | 0
  25 ml/h: number analyzed (Participants) | 0 | 18 | 0
  25 ml/h: number analyzed (Local TEAEs) | 0 | 20 | 0
  25 ml/h |  | 1.2 (0.37) |
  50 ml/h: number analyzed (Participants) | 0 | 14 | 0
  50 ml/h: number analyzed (Local TEAEs) | 0 | 8 | 0
  50 ml/h |  | 1.6 (0.92) |
  75 ml/h: number analyzed (Participants) | 0 | 13 | 0
  75 ml/h: number analyzed (Local TEAEs) | 0 | 2 | 0
  75 ml/h |  | 1.0 (0.00) |
  100 ml/h: number analyzed (Participants) | 0 | 12 | 0
  100 ml/h: number analyzed (Local TEAEs) | 0 | 1 | 0
  100 ml/h |  | 1.0 (NA) — Not estimable because events = 1 |
  30 ml/h: number analyzed (Participants) | 0 | 0 | 16
  30 ml/h: number analyzed (Local TEAEs) | 0 | 0 | 6
  30 ml/h |  |  | 2.2 (2.86)
  60 ml/h: number analyzed (Participants) | 0 | 0 | 16
  60 ml/h: number analyzed (Local TEAEs) | 0 | 0 | 17
  60 ml/h |  |  | 5.6 (12.91)
  120 ml/h: number analyzed (Participants) | 0 | 0 | 14
  120 ml/h: number analyzed (Local TEAEs) | 0 | 0 | 5
  120 ml/h |  |  | 3.0 (2.12)

7. Secondary Outcome: Tolerability of Infusions
Description: Tolerability = number of infusions without severe local adverse events / total number of infusions. Severe = A type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Only events are included which start prior to subject's start date of non-response.
Time Frame: At the end of 4 weeks for each planned infusion parameter
Population: SAS
Measure: Number; unit: Ratio
Units Other Than Participants: Infusions
Arm/Group | IgPro20 (Pump-Assisted Volume Cohort) | IgPro20 (Pump Assisted Flow Rate Cohort) | IgPro20 (Manual Push Flow Rate Cohort)
Number analyzed (Participants) | 15 | 18 | 16
Number analyzed (Infusions) | 152 | 222 | 626
Ratio
  25 ml: number analyzed (Participants) | 15 | 0 | 0
  25 ml: number analyzed (Infusions) | 60 | 0 | 0
  25 ml | 1.00 |  |
  40 ml: number analyzed (Participants) | 12 | 0 | 0
  40 ml: number analyzed (Infusions) | 48 | 0 | 0
  40 ml | 1.00 |  |
  50 ml: number analyzed (Participants) | 11 | 0 | 0
  50 ml: number analyzed (Infusions) | 44 | 0 | 0
  50 ml | 1.00 |  |
  25 ml/h: number analyzed (Participants) | 0 | 18 | 0
  25 ml/h: number analyzed (Infusions) | 0 | 70 | 0
  25 ml/h |  | 1.00 |
  50 ml/h: number analyzed (Participants) | 0 | 14 | 0
  50 ml/h: number analyzed (Infusions) | 0 | 55 | 0
  50 ml/h |  | 1.00 |
  75 ml/h: number analyzed (Participants) | 0 | 13 | 0
  75 ml/h: number analyzed (Infusions) | 0 | 50 | 0
  75 ml/h |  | 1.00 |
  100 ml/h: number analyzed (Participants) | 0 | 12 | 0
  100 ml/h: number analyzed (Infusions) | 0 | 47 | 0
  100 ml/h |  | 0.98 |
  30 ml/h: number analyzed (Participants) | 0 | 0 | 16
  30 ml/h: number analyzed (Infusions) | 0 | 0 | 220
  30 ml/h |  |  | 1.00
  60 ml/h: number analyzed (Participants) | 0 | 0 | 16
  60 ml/h: number analyzed (Infusions) | 0 | 0 | 208
  60 ml/h |  |  | 1.00
  120 ml/h: number analyzed (Participants) | 0 | 0 | 14
  120 ml/h: number analyzed (Infusions) | 0 | 0 | 198
  120 ml/h |  |  | 1.00

ADVERSE EVENTS:
Time Frame: Up to 17 weeks per participant
Groups:
- IgPro20 (Pump-assisted Volume) 25 mL: Volumes per injection site of 25 mL administered subcutaneously.
- IgPro20 (Pump-assisted Volume) 40 mL: Volumes per injection site of 40 mL administered subcutaneously.
- IgPro20 (Pump-assisted Volume) 50 mL: Volumes per injection site of 50 mL administered subcutaneously.
- IgPro20 (Pump-assisted Flow Rate) 25 mL/h: Flow rates per injection site of 25 mL/hour administered subcutaneously.
- IgPro20 (Pump-assisted Flow Rate) 50 mL/h: Flow rates per injection site of 50 mL/hour administered subcutaneously.
- IgPro20 (Pump-assisted Flow Rate) 75 mL/h: Flow rates per injection site of 75 mL/hour administered subcutaneously.
- IgPro20 (Pump-assisted Flow Rate) 100 mL/h: Flow rates per injection site of 100 mL/hour administered subcutaneously.
- IgPro20 (Manual Push Flow Rate) 30 mL/h: Flow rates per injection site of approximately 30 mL/hour administered subcutaneously.
- IgPro20 (Manual Push Flow Rate) 60 mL/h: Flow rates per injection site of approximately 60 mL/hour administered subcutaneously.
- IgPro20 (Manual Push Flow Rate) 120 mL/h: Flow rates per injection site of approximately 120 mL/hour administered subcutaneously.
Arm/Group | IgPro20 (Pump-assisted Volume) 25 mL | IgPro20 (Pump-assisted Volume) 40 mL | IgPro20 (Pump-assisted Volume) 50 mL | IgPro20 (Pump-assisted Flow Rate) 25 mL/h | IgPro20 (Pump-assisted Flow Rate) 50 mL/h | IgPro20 (Pump-assisted Flow Rate) 75 mL/h | IgPro20 (Pump-assisted Flow Rate) 100 mL/h | IgPro20 (Manual Push Flow Rate) 30 mL/h | IgPro20 (Manual Push Flow Rate) 60 mL/h | IgPro20 (Manual Push Flow Rate) 120 mL/h
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12 | 0/11 | 0/18 | 0/14 | 0/13 | 0/12 | 0/16 | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/11 | 0/18 | 0/14 | 0/13 | 0/12 | 0/16 | 1/16 | 0/14
Other Adverse Events (participants affected / at risk) | 4/15 | 4/12 | 1/11 | 7/18 | 4/14 | 3/13 | 3/12 | 5/16 | 8/16 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (Pump-assisted Volume) 25 mL (N=15) | IgPro20 (Pump-assisted Volume) 40 mL (N=12) | IgPro20 (Pump-assisted Volume) 50 mL (N=11) | IgPro20 (Pump-assisted Flow Rate) 25 mL/h (N=18) | IgPro20 (Pump-assisted Flow Rate) 50 mL/h (N=14) | IgPro20 (Pump-assisted Flow Rate) 75 mL/h (N=13) | IgPro20 (Pump-assisted Flow Rate) 100 mL/h (N=12) | IgPro20 (Manual Push Flow Rate) 30 mL/h (N=16) | IgPro20 (Manual Push Flow Rate) 60 mL/h (N=16) | IgPro20 (Manual Push Flow Rate) 120 mL/h (N=14)
suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (Pump-assisted Volume) 25 mL (N=15) | IgPro20 (Pump-assisted Volume) 40 mL (N=12) | IgPro20 (Pump-assisted Volume) 50 mL (N=11) | IgPro20 (Pump-assisted Flow Rate) 25 mL/h (N=18) | IgPro20 (Pump-assisted Flow Rate) 50 mL/h (N=14) | IgPro20 (Pump-assisted Flow Rate) 75 mL/h (N=13) | IgPro20 (Pump-assisted Flow Rate) 100 mL/h (N=12) | IgPro20 (Manual Push Flow Rate) 30 mL/h (N=16) | IgPro20 (Manual Push Flow Rate) 60 mL/h (N=16) | IgPro20 (Manual Push Flow Rate) 120 mL/h (N=14)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 1 (4) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 1 (2) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Injection site pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (7) | 2 (5) | 0 (0) | 1 (1) | 1 (4) | 2 (4) | 1 (1)
Injection site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Injection site discoloration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait inability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT03033745/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03033745/SAP_001.pdf